CLINICAL TRIAL: NCT02431091
Title: Evaluation of the Role of Optical Coherence Tomography (OCT) in the Detection of HIV-associated Neurocognitive Disorder
Brief Title: Evaluation of the Role of OCT in the Detection of HIV-associated Neurocognitive Disorder
Acronym: OCT-HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Fonds iris-Recherche, Fondation Roi Baudouin, Belgium (Unknown)
Responsible Party: Principal Investigator, Agnès Libois, Chef de Clinique, Centre Hospitalier Universitaire Saint Pierre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUSTP-OCTHIV
Record Dates: First submitted 2015-04-22; First posted 2015-04-30 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: AIDS-Related Dementia Complex
Keywords: Optical Coherence Tomography
MeSH Terms: conditions — AIDS Dementia Complex | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Definite Case (Experimental): Patients with abnormal response on both the screening questions and at least one of the cognitive screening tests.
  Optical Coherence Tomography is performed in all definite cases
  Interventions: Other: Optical Coherence Tomography
- Control (Active Comparator): Patients with normal response on both the screening questions and all the cognitive screening tests.
  Optical Coherence Tomography is performed in matched control A patients
  Interventions: Other: Optical Coherence Tomography

INTERVENTIONS:
Other: Optical Coherence Tomography — Optical Coherence Tomography provides a non invasive evaluation of the thickness of different layers of the retina

SUMMARY:
The purpose of this study is to determine the sensitivity and specificity of the use of optical coherence tomography to detect HIV-associated neurocognitive disorder compared to MRI and usual cognitive screening tools.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Antiretroviral treatment
* Undetectable plasmatic HIV viral load (viral load<50 copies/ml) for at least 6 months
* Ability to understand and give approved consent

Exclusion Criteria:

* Any present or past ophthalmologic illness that may impair OCT results
* Previous cerebral infection with sequel
* Previous cerebrovascular disease with sequel
* Severe psychiatric illness
* Active alcohol or drug abuse
* Active chronic hepatitis C
* Inability to perform french cognitive assessment
* Inability to perform a MRI
* Inability to perform a lumbar puncture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal OCT (retinal thickness in µm) in patients with abnormal full neurocognitive evaluation | Baseline

SECONDARY OUTCOMES:
Number of patients with abnormal neuroscreen and/or modified dementia scale in patients with abnoraml full neurocognitve evaluation | Baseline
Correlation between retinal thickness (in µm) and cerebral atrophy in % of brain parenchymal fraction ( measured by cerebral MRI) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Dewit, PhD, Study Director — CHU St Pierre, Service des Maladies Infectieuses
Locations (1):
- Hopital St Pierre, Brussels, Belgium